CLINICAL TRIAL: NCT03592082
Title: Can Use of Bismuth Subsalicylate in Clostridium Difficile Patients Decrease the Length of Stay and Time to Resolution of Symptoms
Brief Title: Use of Bismuth Subsalicylate in Clostridium Difficile Colitis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: Bassett Healthcare (Other)
Responsible Party: Principal Investigator, Jennifer Victory, RN, CCRC, Clinical Research Nurse Supervisor, Bassett Healthcare
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2089
Record Dates: First submitted 2018-01-17; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections | interventions — bismuth subsalicylate

STUDY DESIGN:
Masking Description: none - open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care alone (Active Comparator): Participants will receive standard antibiotic therapy for Clostridium Difficile (CDiff) infection without additional adjuvant therapy.
  Interventions: Drug: standard antibiotic therapy
- Standard care with Bismuth subsalicylate (BSS) (Experimental): Participants will receive BSS524 mg ((2) 262 mg tablets) four times per day for 14 days in addition to standard antibiotic therapy.
  Interventions: Drug: Bismuth Subsalicylate

INTERVENTIONS:
Drug: Bismuth Subsalicylate — BSS 524 mg ((2) 262 mg tablets) given four times per day for 14 days
  Arms: Standard care with Bismuth subsalicylate (BSS)
Drug: standard antibiotic therapy — antibiotic therapy administered per standard protocol
  Arms: Standard care alone

SUMMARY:
Clostridium difficle infection is the leading cause of hospital acquired infection and infectious diarrhea in hospitalized patients. Eradication treatment for this infection is the challenging tasks for clinicians due to treatment resistance developed from new hypervirulent strains. The recurrence rate of this infection is around 20% and there is high likelihood(60-70%) of another episode after index recurrence. Given constant challenge new treatment options are under study. Aim of the study is to evaluate if use of bismuth subsalicylate (BSS) can decrease the length of stay in patients admitted with Clostridium difficile infection. Secondarily investigators will also see if there is any impact of BSS in decrease the recurrence.

DETAILED DESCRIPTION:
Clostridium difficile (C.Diff) infection is the leading cause of hospital acquired infection and infectious diarrhea in hospitalized patients. Eradication treatment for this infection is the challenging task for clinicians due to treatment resistance developed from new hypervirulent strains. The recurrence rate of this infection is around 20% and there is high likelihood (60-70%) of another episode after index recurrence. Given constant challenges new treatment options are under study.

The purpose of this study is to examine if the addition of bismuth subsalicylate (BSS) (the active ingredient in Pepto-Bismol) 524 mg ((2) 262 mg tablets) given four times per day for 14 days to standard of care treatment of C.Diff will decrease the length of stay and decrease the time to resolution of C.Diff symptoms compared to patients who received standard of care treatment for C.Diff alone.

Bismuth subsalicylate has been used for long time in infectious diarrhea and is over the counter drug with few side effects. Studies in hamsters have shown bismuth subsalicylate to be effective in treating C.Diff. Investigators believe given cheaper cost and less side effect profile this drug is worth looking for treatment of C.Diff infection which has a huge burden on health care.

This is an open label, randomized, controlled trial. Hospitalized patients aged 18 years or older with positive stool test for C.Diff toxin will be randomized to one of two treatment groups:

Group 1 will receive standard of care treatment for C.Diff alone Group 2 will receive BSS 524 mg four times daily for 14 days along with standard of care treatment Oral antibiotic therapy will be limited to oral vancomycin 125 mg every 6 hours daily which is the standard dose for the treatment of clostridium difficile.

Length of stay and time to resolution of symptoms will be measured and compared between the two treatment groups as primary outcomes. Resolution of symptoms is defined has having < 3 diarrheal episodes in 24 hours. The study will also record episodes of recurrence, defined as the reappearance of symptoms within 8 weeks of the completion of antibiotic treatment and the resolution of initial symptoms. Recurrence rates will be compared between the two treatment groups as a secondary outcome.

Both Groups 1 & 2 will have 2 week and 8 week follow up phone calls. Group 1 participants will be called 2 weeks after consent/enrollment in the study to verify antibiotic therapy is completed, verify when/if CDiff symptoms resolved, collect data about any adverse events. Group 2 participants will be called 2 weeks after the initiation of study drug (which should be < 24 hours after consent). The visit window will start on the day the participant is scheduled to complete study drug. The purpose of the call will be to verify that both antibiotics and study drug have been completed, verify when/if CDiff symptoms resolved, and collect data about any adverse events.

Both Groups 1 and 2 participants will be called 8 weeks after the expected (or known) completion date of antibiotic therapy prescribed for the treatment of CDiff to see if CDiff symptoms have recurred and if there have been any adverse events..

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Hospitalized patient with documented positive stool test for CDiff
* Able and willing to provide informed consent

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Known allergy to BSS or other salicylates, including aspirin
* History of bleeding disorder
* History of gastrointestinal bleed,
* History of gastrointestinal ulcer
* Chronic use of anticoagulants
* Chronic NSAID use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Length of stay | 70 days (study period = 14 days of antibiotic treatment plus 8 weeks/56 days post treament completion)
  number of days hospitalized after the initiation of treatment for CDiff

SECONDARY OUTCOMES:
Time to resolution of symptoms | 70 days
  Resolution of symptoms is defined as having < 3 diarrheal episodes in 24 hours
CDiff Recurrence | 70 days
  Recurrence is defined as the reappearance of symptoms within 8 weeks of the completion of antibiotic treatment and the resolution of initial symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Abdulhadi Quadri, MD, Principal Investigator — Bassett Medical Center
Locations (1):
- Bassett Healthcare Network, Cooperstown, New York, United States

IPD SHARING:
Plan to Share IPD: No